CLINICAL TRIAL: NCT04606446
Title: A PHASE 1/2A DOSE ESCALATION AND EXPANSION STUDY TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETIC, PHARMACODYNAMIC, AND ANTI-TUMOR ACTIVITY OF PF-07248144 IN PARTICIPANTS WITH ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: Study of PF-07248144 in Advanced or Metastatic Solid Tumors
Acronym: KAT6
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4551001; NCT04606446 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2020-10-05; First posted 2020-10-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic ER+ HER2- Breast Cancer; Locally Advanced or Metastatic Castration-resistant Prostate Cancer; Locally Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: Solid tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fulvestrant; Letrozole; palbociclib

STUDY DESIGN:
Intervention Model Description: The dose escalation parts and the dose finding parts of the study will be guided by a Bayesian analysis of Cycle 1 dose-limiting toxicity (DLT) data for PF-07248144 as monotherapy or in combination (Part 1B, Part 1C, Part 1D and Part 1E).
  A traditional 2-parameter Bayesian Logistic Regression Model (BLRM) will be used to model the DLT relationship of PF-07248144 monotherapy and a more complex BLRM model specifically designed for combinations will be used to model the dose/DLT relationship of PF-07248144 given in combination with fulvestrant, with letrozole + palbociclib, with PF-07220060 + fulvestrant or with vepdegestrant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 1A Monotherapy Dose Escalation (Experimental): PF-07248144 Monotherapy Escalation
  Interventions: Drug: PF-07248144
- 1B Combination Dose Escalation (Experimental): PF-07248144 with Fulvestrant Combination Dose Escalation
  Interventions: Drug: PF-07248144; Drug: Fulvestrant
- 1C Combination Dose Escalation (Experimental): PF-07248144 with Letrozole + Palbociclib Combination Dose Escalation
  Interventions: Drug: PF-07248144; Drug: Letrozole; Drug: Palbociclib
- 2A Monotherapy Dose Expansion Arm (Experimental): PF-07248144 Monotherapy Dose Expansion
  Interventions: Drug: PF-07248144
- 2B Combination Dose Expansion Arm (Experimental): PF-07248144 with Fulvestrant Dose Expansion
  Interventions: Drug: PF-07248144; Drug: Fulvestrant
- 1D Combination Dose Escalation (Experimental): PF-07248144 with PF-07220060 +Fulvestrant
  Interventions: Drug: PF-07248144; Drug: Fulvestrant; Drug: PF-07220060
- 2D Combination Dose Expansion Arm (Experimental): PF-07248144 with PF-07220060 +Fulvestrant Dose Expansion
  Interventions: Drug: PF-07248144; Drug: Fulvestrant; Drug: PF-07220060
- China Monotherapy Dose Expansion (Experimental): PF-07248144 Monotherapy Dose Expansion
  Interventions: Drug: PF-07248144
- 1E Combination Dose Escalation (Experimental): PF-07248144 with Vepdegestrant Combination Dose Escalation
  Interventions: Drug: PF-07248144; Drug: PF-07850327, ARV-471, vepdegestrant
- 2E Combination Dose Expansion Arm (Experimental): PF-07248144 with Vepdegestrant Combination Dose Expansion
  Interventions: Drug: PF-07248144; Drug: PF-07850327, ARV-471, vepdegestrant

INTERVENTIONS:
Drug: PF-07248144 — KAT6 Inhibitor
Drug: Fulvestrant — Endocrine Therapy
  Other Names: Faslodex
  Arms: 1B Combination Dose Escalation; 1D Combination Dose Escalation; 2B Combination Dose Expansion Arm; 2D Combination Dose Expansion Arm
Drug: Letrozole — Endocrine Therapy
  Other Names: Femara
  Arms: 1C Combination Dose Escalation
Drug: Palbociclib — CDK4/6 Inhibitor
  Other Names: Ibrance
  Arms: 1C Combination Dose Escalation
Drug: PF-07220060 — CDK4 inhibitor
  Arms: 1D Combination Dose Escalation; 2D Combination Dose Expansion Arm
Drug: PF-07850327, ARV-471, vepdegestrant — PROTAC (PROteolysis Targeting Chimera) ER degrader
  Arms: 1E Combination Dose Escalation; 2E Combination Dose Expansion Arm

SUMMARY:
This is an open-label, multi center study to evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of PF-07248144 and early signs of clinical efficacy of PF-07248144 as a single agent and in combination with other agents

DETAILED DESCRIPTION:
Study has two parts, Part 1 (dose escalation) and Part 2 (dose expansion). Part 1 is divided into Parts 1A, 1B, 1C, 1D and 1E and Part 2 is divided into Parts 2A, 2B, 2D and 2E. In Part 1A, single escalating doses of PF-07248144 alone will be administered to determine the maximum tolerable dose (MTD) and select the recommended dose for expansion (RDE). In Part 1B, 1C, 1D and 1E PF-07248144 will be administered in combination with either fulvestrant (Part 1B); palbociclib + letrozole (Part 1C) or PF-07220060+fulvestrant (Part 1D) or vepdegestrant (Part 1E). After the determination of the monotherapy RDE in Part 1A, PF-07248144 will be evaluated in a dose expansion cohort as a monotherapy in Part 2A.

After determination of the combination RDE from Part 1B, PF-07248144 in combination with fulvestrant, PF-07248144 will be evaluated in a combination dose expansion with fulvestrant in Part 2B. In Part 1C, PF-07248144 in combination with letrozole + palbociclib will be evaluated for dose finding to determine the MTD and RDE for this combination. After determination of the triple combination RDE from Part 1D, PF-07248144 in combination with PF-07220060 + fulvestrant will be evaluated in a combination dose-expansion cohort, Part 2D. After determination of the combination RDE from Part 1E, PF-07248144 in combination with vepdegestrant will be evaluated in a combination dose-expansion cohort, Part 2E.

ELIGIBILITY:
Inclusion Criteria:

* Disease Characteristics - Breast, Prostate, and Lung Cancer
* Part 1A (Monotherapy Dose Escalation) Histological or cytological diagnosis of locally advanced or metastatic ER+HER2- breast cancer, CRPC, or NSCLC that is intolerant or resistant to standard therapy or for which no standard therapy is available.
* Part 1B, Part 1C, Part 1D and Part 1E (Combination Dose Escalation) Histological or cytological diagnosis of locally advanced or metastatic ER+HER2- breast cancer. Participants must have progressed after at least 1 prior line of treatment with an endocrine therapy and CDK4/6 inhibitor in the advanced or metastatic setting.
* Part 2A (ER+HER2- breast cancer 2L+, monotherapy) Histological or cytological diagnosis of locally advanced or metastatic ER+HER2- breast cancer. Participants must have progressed after at least 1 prior line of CDK4/6 inhibitor and 1 line of endocrine therapy.
* Part 2B (ER+HER2- breast cancer 2-4L, combination with fulvestrant) Histological or cytological diagnosis of advanced or metastatic ER+HER2- breast cancer. Participants must have progressive disease after at least 1 prior line of a CDK4/6 inhibitor and at least 1 prior line of endocrine therapy.. Participants must not have received more than 3 prior lines of systemic therapies including up to 1 line of cytotoxic chemotherapy for visceral disease in advanced or metastatic setting; Participants may have but are not required to have prior treatment with fulvestrant.
* Part 2D (ER+HER2- breast cancer 2-4L, combination with PF-07220060 (CDK4i) and fulvestrant):

Histological or cytological diagnosis of advanced or metastatic ER+HER2- breast cancer. Participants must have progressive disease after at least 1 prior line of a CDK4/6 inhibitor and at least 1 prior line of endocrine therapy.

* Participants must have not received more than 3 lines of systemic therapies including up to 1 line of cytotoxic chemotherapy for visceral disease in advanced or metastatic setting; Participants may have but are not required to have prior treatment with fulvestrant.
* Part 2E (ER+HER2- breast cancer 2-4L, combination with vepdegestrant): Histological or cytological diagnosis of advanced or metastatic ER+HER2- breast cancer. Participants must have progressive disease after at least 1 prior line of a CDK4/6 inhibitor and at least 1 prior line of endocrine therapy; Participants must have not received more than 3 lines of systemic therapies including up to 1 line of cytotoxic chemotherapy for visceral disease in advanced or metastatic setting; Participants may have received fulvestrant
* Participants with ER+HER2- advanced or metastatic breast cancer must have documentation of ER-positive tumor (≥1% positive stained cells) based on most recent tumor biopsy utilizing an assay consistent with local standards.
* Participants with ER+HER2- advanced or metastatic breast cancer must have documentation of HER2-negative tumor: HER2-negative tumor is determined as immunohistochemistry score 0/1+ or negative by in situ hybridization (FISH/CISH/SISH/DISH) defined as a HER2/CEP17 ratio <2 or for single probe assessment a HER2 copy number <4.
* Female participants with ER+HER2- advanced or metastatic breast cancer considered to be of childbearing potential (or have tubal ligations only) must be willing to undergo medically induced menopause by treatment with the approved LHRH agonist such as goserelin, leuprolide or equivalent agents to induce chemical menopause.
* Female participants with ER+HER2- advanced or metastatic breast cancer of nonchildbearing potential must meet at least 1 criteria of achieving postmenopausal status.
* Participants must have at least 1 measurable lesion as defined by RECIST version 1.1 that has not been previously irradiated.
* Eastern Cooperative Oncology Group (ECOG) Performance Status PS 0 or 1
* Female or male patients aged ≥ 18 years (Japan ≥ 20 years) (South Korea ≥ 19 years).
* Adequate renal, liver, and bone marrow function.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade 1 except for adverse events (AEs) not constituting a safety risk by investigator judgment.

Exclusion Criteria:

* Unmanageable ascites (limited medical treatment to control ascites is permitted, but all participants with ascites require review by sponsor's medical monitor).
* Participants with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Major surgery, radiation therapy, or systemic anti-cancer therapy within 3 weeks prior to study entry.
* Prior irradiation to >25% of the bone marrow.
* ECG clinically relevant abnormalities (eg, QTc >470 msec, complete LBBB, second/third degree AV block, ST elevation or EKG changes suggesting myocardial infarction or active myocardia ischemia).
* Therapeutic anticoagulation. However, low molecular weight heparin is allowed. Vitamin K antagonists or factor Xa inhibitors may be allowed following discussion with the Sponsor.
* Known or suspected hypersensitivity or severe allergy to active ingredient/excipients of PF-07248144.
* Active inflammatory GI disease, refractory and unresolved chronic diarrhea or previous gastric resection, lap band surgery or other GI conditions and surgeries that may significantly alter the absorption of PF-07248144 tablets. Gastroesophageal reflux disease under treatment is allowed.
* Pregnant or breastfeeding female participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2028-02-03 (Estimated); Study Completion 2029-09-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities in the Dose Escalation Arms. | Up to 29 days
  Dose-limiting toxicities (DLTs)
Safety and Tolerability as assessed by adverse event monitoring for participants enrolled in the Dose Escalation Arms. | Up to 24 months
  Adverse Events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Safety and Tolerability through monitoring of laboratory assessments for participants enrolled in the Dose Escalation Arms. | Up to 24 months
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Safety and Tolerability as assessed by adverse event monitoring for participants enrolled in the Dose Expansion Arms | Up to 24 months
  Adverse Events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Safety and Tolerability through monitoring of laboratory assessments for participants enroled in the Dose Expansion Arms | Up to 24 months
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.

SECONDARY OUTCOMES:
Single Dose: Maximum Observed Concentration (Cmax) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Single Dose: Time to Maximum concentration (Tmax) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Single Dose: AUC from time zero to time of last measurable concentration (AUClast) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Single and Multiple Dose: Terminal Elimination half-life (t1/2) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Multiple Dose: Steady-State Cmax (Cmax,ss) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Multiple Dose: Steady-state Tmax (Tmax,ss) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Multiple Dose: Steady state AUC during a dosage interval (τ) (AUCτ,ss) in the Dose Escalation and Dose Finding Arms | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Multiple Dose: Steady-state Cmin (Cmin,ss) in the Dose Escalation and Dose Finding Arms. | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Multiple Dose: Steady-state apparent total clearance (CLss/F) in the Dose Escalation and Dose Finding Arms. | Up to 24 months
  Pharmacokinetic (PK) assessments for PF-07248144, PF-07220060 (Part 1D) and vepdegestrant and ARV-473 (Part 1E)
Palbociclib trough concentrations at steady instate (Cmin,ss) in the 1C combination dose finding arm. | Up to 24 months
  Pharmacokinetic (PK) assessment for palbociclib exposure.
Peak concentrations of PF-07248144, PF-07220060 (Part 2D) and vepdegestrant and ARV-473 (Part 2E) for selected cycles in the Dose Expansion Arms | Up to 24 months
  Pharmacokinetic (PK) assessment for PF-07248144, PF-07220060 (Part 2D) and vepdegestrant and ARV-473 (Part 2E)
Trough concentrations of PF-07248144 for selected cycles in the Dose Expansion Arms | Up to 24 months
  Pharmacokinetic (PK) assessment for PF-07248144 , PF-07220060 (Part 2D) and vepdegestrant and ARV-473 (Part 2E)
Maximum Observed Concentration (Cmax) in the participants in the food effect subset in monotherapy dose expansion arm | Cycle 1 Day -7 and Cycle 1 Day 1 (each cycle is 28 days)
  The effect of food on the PK of PF-07248144.
Time to Maximum concentration (Tmax) in the participants in the food effect subset in monotherapy dose expansion arm | Cycle 1 Day -7 and Cycle 1 Day 1 (each cycle is 28 days)
  The effect of food on the PK of PF-07248144.
AUC from time zero to time of last measurable concentration (AUClast) in the participants in the food effect subset in monotherapy dose expansion arm | Cycle 1 Day -7 and Cycle 1 Day 1 (each cycle is 28 days)
  The effect of food on the PK of PF 07248144.
Amount of PF-07248144 excreted in urine relative to dose administered (%) in a sub-set of participants in monotherapy dose expansion arm. | Up to 24 months
  Evaluate urine pharmacokinetic (PK) of PF-07248144.
Renal clearance (CLr) in a sub-set of participants in monotherapy dose expansion arm | Up to 24 months
  Evaluate urine pharmacokinetic (PK) of PF-07248144.
Progression Free Survival (PFS) observed in participants in the Dose Expansion Arms | Up to 24 months
Time to Progression (TTP) observed in participants enrolled in the Dose Expansion Arms | Up to 24 months
Overall survival (OS) observed in participants enrolled in Dose Expansion Arms | Up to 24 months
Best Overall Response (BOR) observed in participants in the dose expansion arms | Up to 24 months
Duration of Response (DOR) observed in participants in the dose expansion arms | up to 24 months
Clinical Benefit Rate (CBR) observed in participants in the Dose Expansion Arms | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (20):
  - HonorHealth, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Cedars-Sinai Medical Center; SOCCI Pharmacy, Los Angeles, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Smilow Cancer Hospital at Yale - New Haven, New Haven, Connecticut
  - Yale-New Haven Hospital- Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University Medical Center, lnc.:DBA University of Louisville Hospital, Louisville, Kentucky
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute / Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (6):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Western Health-Sunshine & Footscray Hospitals, St Albans, Victoria
  - St. John of God Subiaco Hospital, Subiaco, Western Australia
- China (5):
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
- Japan (4):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa cancer center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam, Ky?nggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-kwangyǒkshi
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Mukohara T, Park YH, Sommerhalder D, Yonemori K, Hamilton E, Kim SB, Kim JH, Iwata H, Yamashita T, Layman RM, Mita M, Clay T, Chae YS, Oakman C, Yan F, Kim GM, Im SA, Lindeman GJ, Rugo HS, Liyanage M, Saul M, Le Corre C, Skoura A, Liu L, Li M, LoRusso PM. Inhibition of lysine acetyltransferase KAT6 in ER+HER2- metastatic breast cancer: a phase 1 trial. Nat Med. 2024 Aug;30(8):2242-2250. doi: 10.1038/s41591-024-03060-0. Epub 2024 Jun 1. PMID 38824244
- [Derived] Bishop TR, Subramanian C, Bilotta EM, Garnar-Wortzel L, Ramos AR, Zhang Y, Asiaban JN, Ott CJ, Rock CO, Erb MA. Acetyl-CoA biosynthesis drives resistance to histone acetyltransferase inhibition. Nat Chem Biol. 2023 Oct;19(10):1215-1222. doi: 10.1038/s41589-023-01320-7. Epub 2023 May 1. PMID 37127754
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4551001